CLINICAL TRIAL: NCT05619419
Title: Feasibility and Efficacy of a Mindfulness-enhanced Positive Affect Induction for Experimentally Induced Pain
Brief Title: Study of Affect Induction for Lab Induced Pain in Healthy Undergraduates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: 20-0030
Record Dates: First submitted 2022-10-20; First posted 2022-11-16 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Meditation; Pain; Mindfulness; Affect; Emotion Regulation
Keywords: Mindfulness-enhanced; Positive affect; Meditation; Pain self-management; Behavioral; Mindfulness; Mindfulness-enhanced positive affect induction (MPAI); Experimentally induced pain; Cold pressor test (CPT); Breathing Meditation (BM); Natural Response (NR)
MeSH Terms: conditions — Pain; Emotional Regulation; Behavior

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of three groups: mindfulness-enhanced positive affect induction (MPAI), breathing meditation (BM), or natural response (NR). Pain will be induced via a cold pressor test (CPT), as the CPT can closely resemble tonic increasing pain similar to that of pain flares. Participants will be instructed to either respond naturally, use the MPAI, or breathing meditation for managing pain during the CPT. Relevant pain related outcomes and covariates will be assessed via baseline and post-CPT questionnaires. The MPAI is the primary intervention being examined, with the BM and NR groups as active comparison and control groups respectively.
Masking Description: Research assistant will be aware of participant randomization, as necessary for providing the correct study instructions and procedures (e.g., pain psycho-education and meditation audio recording). Participants will not be masked, as they will receive specific instructions on and audio recorded meditation practice based on their group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mindfulness-enhanced positive affect induction (MPAI) (Experimental): The MPAI is a method of bringing mindful (nonjudgmental) awareness to positive emotions, thoughts, and memories and is not expected to result in adverse experiences. It includes beginning with mindful awareness of the breath (i.e., meditation focusing on the breath) to draw attention away from negative aspects of pain. With continued awareness of the breath, smiling and gentle laughter are begun in order to initiate positive affect. With continued smiling and laughter, participants then imagine the smiles and laughter of those they are fond of, to allow a positive affect state to build upon itself and trigger state dependent positive memories, thoughts, emotions (e.g., gratitude) and self-efficacy of pain management.
  Interventions: Behavioral: Mindfulness-enhanced positive affect induction
- Breathing meditation (BM) (Active Comparator): Breathing meditation is a method of bringing mindful (nonjudgmental) awareness to various aspects of the breath and is aimed toward attaining a neutral state of affect and is not expected to result in adverse experiences. It involves bringing present-moment focused, nonjudgmental awareness to aspects breathing, such as sensations of airflow with each inhalation and exhalation, as well noticing the rise and expansion of the chest and belly with each inhalation. The use of breathing mediation will serve as a comparison task for the MPAI.
  Interventions: Behavioral: Breathing Meditation
- Natural Response (NR) (No Intervention): Participants instructed to respond naturally to the cold pressor test will be instructed to not attempt to modify or control their experience (e.g., via distraction or use of meditation). Natural response will serve as a control comparator for the MPAI and is not expected to result in adverse experiences.

INTERVENTIONS:
Behavioral: Mindfulness-enhanced positive affect induction — Participants will receive brief psychoeducation about biopsychosocial pain management and practice with the MPAI via guided audio recording. They will then listen to the audio recording a final time before beginning the cold pressor test for experimental pain induction. They will be instructed to continue using the MPAI to manage pain during the cold pressor test.
  Other Names: MPAI
  Arms: Mindfulness-enhanced positive affect induction (MPAI)
Behavioral: Breathing Meditation — Participants will receive brief psychoeducation about biopsychosocial pain management and practice with the BM via guided audio recording. They will then listen to the audio recording a final time before beginning the cold pressor test for experimental pain induction. They will be instructed to continue using the BM to manage pain during the cold pressor test.
  Other Names: BM
  Arms: Breathing meditation (BM)

SUMMARY:
The goal of this clinical trial is to test if a mindfulness-enhanced positive affect induction (MPAI) works well to reduce pain intensity and pain unpleasantness from a cold water pain test in undergraduate college students who do not endorse ongoing medical or mental health diagnoses. The main questions it aims to answer are:

* Is the MPAI a feasible and acceptable psychological technique for managing brief pain?
* Does the MPAI work well to reduce pain intensity and unpleasantness from experimentally induced brief pain, compared to those using a breathing meditation or those instructed to respond naturally.
* Does using the MPAI work well to improve confidence in self-managing brief pain?

Participants will be asked to complete questionnaires about their sleep, pain beliefs, and emotions after consenting to participate and at the end of the study session. They will then be randomized to either:

* Use the MPAI for managing pain induced by a cold water test (placing their hand in a container of cold water kept at approximately 5 degrees Celsius).
* Use a breathing meditation for managing pain induced by a cold water test (placing their hand in a container of cold water kept at approximately 5 degrees Celsius).
* Respond naturally to pain induced by a cold water test (placing their hand in a container of cold water kept at approximately 5 degrees Celsius).

Researchers will compare the MPAI group to the breathing meditation and natural response groups to see if the MPAI group reports less pain from the cold water test and

DETAILED DESCRIPTION:
The purpose of the study is to assess the following aims:

Aim 1: Examine the feasibility and acceptability of a mindfulness-enhanced positive affect induction (MPAI) for improving the experience of experimentally-induced pain.

Aim 2: Examine the efficacy of the MPAI in reducing pain intensity and increasing pain tolerance.

Aim 3: Examine change in self-efficacy in pain management from before and after using the MPAI.

Recruitment:

Participants will be recruited via the University of Colorado (CU) Denver Psychology Participant Pool website (Sona system), a resource for undergraduate Psychology students to participate in research projects. Interested participants will be provided inclusion/exclusion criteria and instructed to register for a study session only if they meet those criteria. Inclusion/exclusion criteria will be confirmed by study research assistants (RAs) during the informed consent process. Participants will receive course credit for participation in the study. If students do not wish to participate in the study, an alternative assignment will be available for equal credit.

The target population will consist of a convenience sample of healthy undergraduate students at CU Denver. While this population does not generalize to populations with chronic pain, as this is the first study of this particular affect induction for pain, the primary goal is to assess general feasibility and efficacy, which may influence future research specific to chronic pain populations. The population will be randomized into three experimental groups: MPAI, breathing meditation (BM), and natural response (NR). The BM and NR groups will serve active comparison and control groups respectively. Each group will consist of 46 participants (N=138) based on power analyses accounting for medium effects found in similar studies. Final power analyses were conducted for planned ANCOVAs with f = 0.27, alpha = 0.05, and power = 0.80.

Phone screening will occur in instances in which participants contact study personnel via methods other than CU Denver's Sona system (e.g., via phone or email). Screening questions will not go beyond inclusion criteria listed on an approved study advertisement. No information will be recorded on specific inclusion/exclusion criteria met. Additionally, participants do not provide specific medical details during the consent process. Participants only indicate if they do or do not meet all inclusion/exclusion criteria.

Study Procedures:

Participants will come into the laboratory, provide informed consent, be randomized to one of three groups (natural response, breathing meditation, or positive affect induction) and will complete forms and questionnaires on demographics, sleep quality, positive and negative affect, present-moment affect, pain catastrophizing, mood states (e.g., anger and fatigue), present-moment anxiety, and self-efficacy of pain management. Participants will then receive instructions and practice for their randomized group assignment (e.g., on how to use the positive affect induction). Participants will then complete a cold pressor task (CPT) while using the strategy they were instructed to use (i.e., naturally responding, using breathing meditation, or using the positive affect induction). Importantly, participants will be instructed to begin with their strategy 5 minutes prior to beginning the CPT, to ensure the strategy may have an effect during the CPT, which has a maximum duration of 5 minutes. Participants will then complete a final brief questionnaire rating their pain intensity, pain unpleasantness, present moment affect, self-efficacy of pain management, and feasibility and acceptability of the strategy used.

The CPT is an acute pain task wherein participants put their hand in a cold-water bath. Ice packs will be used within the water bucket to maintain a temperature no greater than 41.0 degrees Fahrenheit (5 degrees Celsius), and participants will have their hand in the water for no greater than five minutes (a maximum time limit of five minutes will be set to prevent any adverse, hypothermic effects from the cold water). The participant will provide both subjective (self-report pain intensity and unpleasantness) and objective (observation of/timed contact with water) measures from the acute pain task. Self-report measures will be taken directly following the CPT. Pain tolerance will be measured via timing when participants remove their hand from the water. The participants will be timed for how long they keep their hand in the water (observation of contact).

Data Collection & Management:

Electronic case report forms and study data management will be performed using the REDCap Study Data Management System through the Colorado Clinical and Translational Sciences Institute (CCTSI) Informatics Core. REDCap is a HIPAA-compliant research data management system developed at Vanderbilt University and deployed at over 1500 institutions. At CU Denver-Anschutz, REDCap is supported by the Office of Information Technology's Development and Informatics Service Center (DISC) and the CCTSI Informatics Core. The CU Denver REDCap installation has passed a rigorous 6-week security threat analysis performed by the CU Denver-Anschutz HIPAA Security Officer. All study data are stored on a secure database server which is separate from the web-facing server -- a best-practices for internet-based security. All user access requires unique user accounts and passwords. All user actions are recorded in a secure audit log. The database server is routinely backed-up. All security patches and application updates are applied immediately upon release by DISC.

Unanticipated Problems/Adverse Events Reporting:

Unanticipated problems and adverse events will be reported to the Colorado Multiple Institutional Review Board within 5 days of an event.

Statistical Analysis Plan:

Data quality checks will be performed to ensure data included in analyses are interpretable, consistent, and within range.

Manipulation Checks:

To assess whether the affect induction and breathing meditation increase positive affect, paired t-tests will be conducted on present-moment affect measures from baseline and post-CPT questionnaires.

Aim 1 To assess feasibility, a one-way ANOVA will be run between groups as a manipulation check for MPAI efficacy. Means, standard deviations, and percentages will additionally be calculated for feasibility and acceptability items. Good feasibility and acceptability will be considered by an a priori threshold of high participant mean ratings (≥80%) for each item.

Aim 2 To assess efficacy of the MPAI on pain from the CPT, one-way ANCOVAs will be calculated to analyze omnibus between-group effects for each pain measure (i.e., for CPT pain tolerance, intensity, and unpleasantness). Post-hoc comparisons will then be calculated to determine specific group differences (e.g., PA vs BM, PA vs NR, and BM vs NR). Correlation analyses will be run on all covariates, to assess for multicollinearity prior to inclusion in ANCOVA analyses. Covariates to be analyzed include: Patient Reported Outcomes Measurement Information System (PROMIS) sleep disturbance (past seven days), PANAS (positive and negative affect past seven days), baseline present-moment affect, pain catastrophizing, present-moment anxiety, baseline PBQ (self-efficacy of pain management), gender, and meditation experience.

Aim 3 To assess for change in self-efficacy in pain management, a paired t-test will be calculated between baseline and post-CPT PBQ scores. A linear mixed model will additionally be calculated to assess change differences between groups; however, as the primary goal of Aim 3 is not to assess between group changes in pain management self-efficacy, this will be an exploratory analysis.

Study Hypotheses:

Aim1. Hypothesis 1. It is hypothesized that the mindfulness-enhanced positive affect induction will have good feasibility and acceptability for improving the experience of experimentally induced pain, based on an a priori threshold of ≥80% mean ratings on related measures.

Aim 2. Hypothesis 1. Compared to the BM and NR groups, the MPAI will result in significantly greater pain tolerance, less pain intensity, and less pain unpleasantness in relation to the experimentally induced pain.

Aim 3. Hypothesis 1. Self-efficacy in pain management will significantly increase from baseline to post-CPT, for the MPAI and BM groups.

Hypothesis 2. A repeated measures ANOVA will show increased PBQ scores for the MPAI and BM groups; however, no changes in PBQ

ELIGIBILITY:
Inclusion Criteria:

* University of Colorado Students
* Age 18-65
* Fluent in written and spoken English

Exclusion Criteria:

* Presence of an untreated mood or psychiatric disorder
* Presence of a current chronic pain condition
* Presence or history of Reynaud's syndrome, peripheral neuropathy, or unstable heart condition (including myocardial infarction, abnormal heart rhythms, or hypertension)
* Current use of prescription pain medication, high-dose anti-psychotics, selective serotonin re-uptake inhibitors (SSRIs), benzodiazepines, or gabapentin
* Day-of over the counter pain medication use
* Marijuana, Cannabidiol (CBD), or psilocybin use within three days of study participation (recency of use assessed via self-report)
* Food, caffeine, and nicotine are not to be had within 30 minutes of cold pressor test (nicotine patch not exclusionary due to stable/consistent state).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2022-11-14 (Actual); Study Completion 2022-11-14 (Actual)

PRIMARY OUTCOMES:
Pain Tolerance, assessed by duration of CPT | Pain tolerance, assessed by duration of the CPT, will be recorded immediately after the intervention (i.e., the CPT), during the post-CPT survey set
  Pain tolerance will be assessed via the amount of time (i.e., number of seconds) until participants remove their hand from the cold water during the cold pressor test (CPT). CPT duration will be timed via a stopwatch and will begin when the participant's hand is submerged in the cold water up to the wrist and will stop immediately when the hand is removed. More time in the water will be indicative of greater pain tolerance. Water temperature will be maintained at 5 degrees Celsius to optimize potential for pain intensity and tolerance during the CPT measures. Longer duration of the CPT will indicate higher pain tolerance.
Pain Intensity, assessed by VAS | Pain intensity will be collected immediately after the intervention (i.e., the CPT) during the post-CPT survey set.
  Pain intensity will be assessed via two items: "Please rate your peak pain intensity experienced during the cold water test" and "Please rate your average pain intensity experienced during the cold water test". Each item response will be rated on a 0-100 visual analog scale (VAS). "0" will indicate no pain intensity and "100" will indicate intolerable pain intensity, with higher scores indicating higher pain intensity.
Pain Unpleasantness, assessed by VAS | Pain unpleasantness will be collected immediately after the intervention (i.e., the CPT) during the post-CPT survey set.
  Pain unpleasantness will be assessed via two items: "Please rate your peak pain unpleasantness experienced during the cold water test (e.g., how bothersome you found the pain from the cold water test)" and "Please rate your average pain unpleasantness experienced during the cold water test (e.g., how bothersome you found the pain from the cold water test)". Each item response will be rated on a 0-100 visual analog scale (VAS). "0" will indicate no pain unpleasantness and "100" will indicate intolerable pain unpleasantness, with higher scores indicating higher pain unpleasantness.
Feasibility beliefs of MPAI as implementable and efficacious for pain management, assessed by three PBQ items | Feasibility measures (i.e., the PBQ) will be collected immediately after the intervention (i.e., the CPT) during the post-CPT survey set.
  Feasibility beliefs of MPAI in pain management will be assessed via three items from the Pain Beliefs Questionnaire (PBQ): "Would you be able to perform the coping strategy while in pain?", 2) "How well will you be able to focus your attention on the coping strategy while in pain?", 3) "How confident are you that you will be able to use the coping strategy to reduce your pain while in pain?". Item responses will be given on a 0-6 seven-point Likert scale with anchors varying by the item (e.g. Not at all Confident/Very Confident, Not at all Well/Very well, and Very Uncertain/Very Certain). Means and percentages will be calculated. Good feasibility with PBQ items will be considered by high mean percentage ratings (≥80%) for each item, with higher mean percentages will indicating greater feasibility (see Outcome 6 below for detail on PBQ). Although the PBQ will be assessed at multiple time points, feasibility analyses will only include items assessed immediately after the intervention.
Acceptability of MPAI as a technique for reducing pain, assessed by six questions on satisfaction and usefulness of the MPAI | Acceptability questions will be assessed immediately after the intervention (i.e., the CPT) during the post-CPT survey set.
  Acceptability will be assessed via the following items: "How acceptable did you find the coping strategy to be?", "How satisfied are you with the coping strategy?", "How useful was the coping strategy?", "Was the coping strategy easy to understand?", "Was the coping strategy easy to use?", "How likely are you to use the coping strategy you learned today?". Item responses will be given on a 0-6 seven-point Likert scale with anchors varying by the item (e.g. Not at all Acceptable/Very Acceptable, Not at all Satisfied/Very Satisfied, Not at all Useful/Very Useful, Extremely Difficult to Understand/Very Easy to Understand, Extremely Difficult to Use/Very Easy to Use, and Not at all Likely/Highly Likely). Means, standard deviations, and percentages of PBQ items will be calculated. Good acceptability will be considered by high mean percentage ratings (≥80%) for each item, with higher mean percentages indicating greater acceptability.
Self-Efficacy in Pain Management assessed by change in Pain Beliefs Questionnaire (PBQ) total scores | Self-efficacy in pain management, assessed by change in PBQ total scores will be assessed during the baseline survey set and the post-CPT survey set (i.e., immediately after the intervention)
  Self-efficacy in pain management will be assessed via the Pain Beliefs Questionnaire (PBQ). The PBQ is a nine-item instrument assessing beliefs in ability to manage pain, as well as ability to learn and utilize a pain self-management technique, with high internal consistency (Chronbach's alpha = 0.89). Example items include: "The degree of pain I experience is mostly up to me" and "How well will you be able to focus your attention on the coping strategy while in pain?". Item responses are given on a 1-7 seven-point scale with anchors such as True/False, Agree/Disagree, Difficult/Easy, Very Little Control/Complete Control, Very Uncertain/Very Certain, Not at all Well/Very well, and Not at all Confident/Very Confident. Total PBQ scores are calculated as the mean of all nine items, with higher scores representing higher levels of self-efficacy in pain management

SECONDARY OUTCOMES:
Present-Moment Affect, assessed by affect ratings | Present-moment affect will be collected during baseline, before the CPT (after condition practice), immediately following the CPT
  Present-moment affect will be assessed via single-item overall affect measures. The purpose for single-item measures is to capture general state affect, which may not be captured via the Positive and Negative Affect Schedule (PANAS). For example, although gratitude is an aspect of positive affect likely to be influenced by the affect induction, it is not an item directly captured with the PANAS. Present-moment affect ratings will be collected to assess manipulation checks of affect induction, as well as influences of present-moment affect on the relationship between affect induction and CPT outcomes. Positive affect will be assessed via the item: "Please rate the extent you currently feel positive emotion". Negative affect will be assessed via the item "Please rate the extent you currently feel negative emotion". Item responses will be rated on a 1-5 five-point scale ranging from "Very slightly or not at all" to "Very much", with higher scores indicating stronger affect.
Positive Affect Manipulation Check | The positive affect manipulation check measure will be assessed pre-intervention [i.e., immediately after practice of the respective meditation, immediately before using the respective meditation during the cold pressor task (CPT)]
  A manipulation check for the positive affect induction will be assessed via a question asking: "Did you experience an increase in positive emotion during the meditation?". If "No" is selected, a follow-up question will prompt participants to select the following relevant factors/reasons, as is appropriate for them: "I am having a bad day/week", "I have experienced a negative life event related to the meditation topic", "I have experienced a negative life event unrelated to the meditation topic", "I am tired/have not slept well recently", "I was not able to focus on the meditation", "I am anxious or fearful about upcoming life events", "I am not in a good mood right now". This will be collected with those randomized to the mindfulness-enhanced positive affect induction (MPAI) and breathing meditation (BM) groups, as part of checking for sufficient practice with their respective meditations.

OTHER OUTCOMES:
Demographics | Demographics will be assessed during the baseline survey set
  A general demographics form will be used to obtain information regarding participant age, gender, race/ethnicity, and socioeconomic status (SES).
Positive and Negative Affect (past 7 days), assessed by PANAS | The PANAS will be assessed during the baseline survey set
  Positive and negative affect from the previous seven days will be assessed via the Positive and Negative Affect Schedule (PANAS). The PANAS assesses overall positive affect (PA) and negative affect (NA) across 20 items (10 positive affect and 10 negative affect), with high internal consistency (0.88 PA, 0.85 NA), convergent validity (.89 - .95) and divergent validity (-.02 - -.18). Temporal instruction will be specific to past week (e.g., "Please indicate the extent to which you have felt this way during the past week"), to assess for the influence of recent affect states on the relationship between affect induction and cold pressor test (CPT) outcomes. Item responses are rated on a 1-4 four-point scale ranging from "very slightly or not at all" to "very much". Example positive affect (PA) items include: enthusiastic, inspired, and interested. Example negative affect (NA) items include: nervous, ashamed, and afraid.
Pain Catastrophizing, assessed by the PCS | The PCS will be assessed during the baseline survey set
  Pain catastrophizing will be assessed via the Pain Catastrophizing Scale (PCS). The PCS assesses negative mental states experienced during or in anticipation of a painful event (e.g., "I feel I can't stand it anymore" and "I can't seem to keep it out of my mind"). The PCS assesses pain catastrophizing across 13 items and three domains (rumination, magnification, and helplessness). It has been shown to have high internal consistency across subscales with alphas of 0.87 (total PCS score), 0.87 (rumination), 0.66 (magnification), and 0.78 (helplessness). As pain catastrophizing has been shown to be associated with numerous pain-related outcomes, it is being collected to assess its influence on the relationship between affect induction and CPT outcomes. Items assess various thoughts surrounding the experience of pain. Item responses are rated on a 0-4 five-point scale, with anchors of "Not at all" to "All the time", with higher scores indicating higher pain catastrophizing.
Sleep Quality (past 7 days), assessed by the SD-sf 8a | The SD-sf 8a will be assessed during the baseline survey set
  Sleep from the past seven days will be assessed via the PROMIS Sleep Disturbance - short form 8a (SD-sf 8a). The SD-sf 8a is a validated measure of sleep disturbance in the past seven days, with conventional reliability of approximately .90 and above for SD-sf-8a. Sleep from the past seven days will be collected to assess the influence of the previous week's sleep quality on the relationship between affect induction and CPT outcomes. Item responses are rated on a 1-5 five-point scale, with anchors ranging from "Not at all" to "Very much", "Never" to "Always", and "Very poor" to "Very good". Example items from the SD-sf 8a include: In the past seven days "My sleep was restless", "I had trouble staying asleep", and "I got enough sleep". Higher scores indicate worse sleep quality.
Mood States, assessed by the POMS-SF | The POMS-SF will be assessed during the baseline survey set
  The profile of mood states - short form (POMS-SF) is a 37-item questionnaire assessing six different mood states: tension, anger, depression, fatigue, vigor, and confusion. Instructions are for respondents to select the number that best describes how they feel "right now". Items are in a checklist format, in which adjectives for each of the six mood states are listed and rated on a 0-4 scale, with 0=Not at all, 1=A little, 2=Moderately, 3=Quite a bit, and 4=Extremely. The POMS-SF has been shown to have good internal consistency with Cronbach's alphas ranging between .76 (confusion) and .95 (depression) across the six mood state categories, as well good convergent validity with correlations of .63 with the Center for Epidemiologic Studies Depression (CES-D) Scale. Higher scores indicate higher intensity of a respective mood state.
Present moment anxiety, assessed by single anxiety rating | Present moment anxiety will be assessed during the baseline survey set
  Present moment anxiety will be assessed via a single-item: "Please rate your current level of anxiety (related or unrelated to the study)". Item responses will be rated on a 1-5 five-point scale with anchors ranging from "None at all" to "Extreme anxiety". Present-moment anxiety will be collected to assess the influence of anxiety on the relationship between affect induction and CPT outcomes. Higher scores indicate higher intensity of anxiety.
Meditation Experience | Meditation experience will be assessed during the baseline survey set
  Meditation experience will be assessed via two items: "How many hours per week do you meditate?" and "Please describe your typical method of meditation". Number of hours per week will be provided via radio buttons ranging from "0" to "10+". Method of meditation will only be assessed if number of hours per week is greater than zero (via REDCap branching logic). Responses to method of meditation will be open-ended via a text box. Meditation experience will be collected to assess the influence of meditation experience on the relationship between affect induction and CPT outcomes, as the affect inductions do involve an aspect of formal meditation (e.g., focusing on the breath, bodily sensations, and emotions).
Handedness | Handedness will be assessed during the baseline survey set
  Handedness will be assessed via a single item: "Please record your handedness". Item responses will include "Right handed", "Left handed", and "Ambidextrous". The purpose of assessing handedness is to ensure the non-dominant hand is used for each CPT.

CONTACTS AND LOCATIONS:
Overall Officials: Dustin S Goerlitz, MA, Principal Investigator — University of Colorado, Denver; Amy Wachholtz, PhD, Study Chair — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
Due to the pilot level nature of the study, we believe it would be inappropriate to allow full open access to the data. If researchers are interested in aspects of the data or would like copies of de-identified data, they may contact the study chair, Dr. Wachholtz.

REFERENCES:
- [Background] Tonelli ME, Wachholtz AB. Meditation-based treatment yielding immediate relief for meditation-naive migraineurs. Pain Manag Nurs. 2014 Mar;15(1):36-40. doi: 10.1016/j.pmn.2012.04.002. Epub 2012 Jun 20. PMID 24602422
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Darnall BD, Sturgeon JA, Kao MC, Hah JM, Mackey SC. From Catastrophizing to Recovery: a pilot study of a single-session treatment for pain catastrophizing. J Pain Res. 2014 Apr 25;7:219-26. doi: 10.2147/JPR.S62329. eCollection 2014. PMID 24851056
- [Background] Mitchell LA, MacDonald RA, Brodie EE. Temperature and the cold pressor test. J Pain. 2004 May;5(4):233-7. doi: 10.1016/j.jpain.2004.03.004. PMID 15162346
- [Background] Rokke PD, al Absi M, Lall R, Oswald K. When does a choice of coping strategies help? The interaction of choice and locus of control. J Behav Med. 1991 Oct;14(5):491-504. doi: 10.1007/BF00845106. PMID 1744911
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] 1. Sullivan MJL, Bishop SR, Pivik J. The Pain Catastrophizing Scale: Development and validation. Psychological Assessment. 2009;7(4):524-532. doi:10.1037/1040-3590.7.4.524
- [Background] Yu L, Buysse DJ, Germain A, Moul DE, Stover A, Dodds NE, Johnston KL, Pilkonis PA. Development of short forms from the PROMIS sleep disturbance and Sleep-Related Impairment item banks. Behav Sleep Med. 2011 Dec 28;10(1):6-24. doi: 10.1080/15402002.2012.636266. PMID 22250775
- [Background] Curran S, Andrykowski M, Studts J. Short Form of the Profile of Mood States (POMS-SF): Psychometric information. Psychological Assessment. Published online March 1995. Accessed January 11, 2020. https://www.academia.edu/1578109/Short_Form_of_the_Profile_of_Mood_States_POMS-SF_Psychometric_information